CLINICAL TRIAL: NCT05983328
Title: A Randomized, Open-label, Single Dose, Crossover Design Phase I Study to Evaluate Tolerability, Safety and Pharmacokinetics of HUYPS-1 in Healthy Volunteers
Brief Title: Phase I Pharmacokinetic Study of HUYPS-1 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinew Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Oral HUYPS-1-001
Record Dates: First submitted 2018-03-05; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-04

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers dose 1 (Experimental): Evaluate tolerability, safety and pharmacokinetic properties of HUYPS-1 after 1 tablet oral administration in healthy subjects
  Interventions: Drug: HUYPS-1 one tablet
- Healthy Volunteer dose 2 (Experimental): Evaluate tolerability, safety and pharmacokinetic properties of HUYPS-1 after 9 tablets oral administration in healthy subjects
  Interventions: Drug: HUYPS-1 nine tablets

INTERVENTIONS:
Drug: HUYPS-1 one tablet — After 7-day washout time, subjects will receive HUYPS-1 1 tablet.
  Arms: Healthy Volunteers dose 1
Drug: HUYPS-1 nine tablets — After 7-day washout time, subjects will receive HUYPS-1 9 tablets.
  Arms: Healthy Volunteer dose 2

SUMMARY:
Fasting Period: At least 10 hours prior to dosing until 4 hours post-dose of each study period.

Period: 24 hours post dose in each period. Each subject will complete two study periods.

Washout Period: At least one week after dosing of the previous period.

Confinement: From at least 10 hours prior to dosing until at least 12 hours post-dose, for a total of at least 22 hours for each study period.

DETAILED DESCRIPTION:
This study is a single center and open-label design to evaluate tolerability, safety and pharmacokinetic properties of HUYPS-1 after single oral administration in healthy subjects under fasting conditions. A total of 14 eligible subjects are expected to be enrolled to ensure 12 evaluable subjects. The study will be completed when there are at least 12 evaluable subjects. The evaluable subjects are those who have completed both periods. Eligible subjects will be randomly assigned to either of the two treatment sequences.

The study design in a 2-sequence, 2-period crossover design. There is at least 7-day washout time between periods. The formulation of HUYPS-1 for oral administration contains 100 mg mannitol and 100 mg sucralose per tablet will be given by one or nine tablets per person of each period. Mannitol and sucralose are both commonly used excipients approved by WHO. These excipients are included in the FDA Inactive Ingredients Guide, GRAS (generally recognized as safe) and commonly used pharmaceutical excipients, therefore the oral doses of these excipients can be regarded as extremely safe in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy adult subjects between 20-50 years of age.
2. Acceptable medical history and physical examination including:
3. Acceptable clinical laboratory determinations without significant deviation from normal values within two months prior to Period I dosing, which includes AST (SGOT), ALT (SGPT), r-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol, triglyceride (TG) and galactose single point (GSP).
4. Acceptable hematology within two months prior to the study, which includes hemoglobin, hematocrit, red blood cells, MCV, MCH, MCHC, white blood cells, differential white blood cells and platelets.
5. Acceptable urinalysis within two months prior to the study, which includes pH, blood, glucose and protein.
6. Signed the written informed consent to participate in this study.
7. Acceptable body mass index (BMI): 18.5 < BMI < 25 kg/m2

Exclusion Criteria:

1. Recent history of drug or alcohol addiction or abuse within the past year.
2. A clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
3. History of allergic response(s) to mannitol, sucralose or related drugs.
4. History of clinically significant allergies including drug allergies or allergic bronchial asthma.
5. Evidence of chronic or acute infectious diseases.
6. Any clinically significant illness or surgery during the one month prior to Period I dosing (as determined by the clinical investigator).
7. Taking any drug known to induce or inhibit hepatic drug metabolism within one month prior to the beginning of the study.
8. Receiving any investigational drug within one month prior to Period I dosing.
9. Taking any prescription medication or any nonprescription medication within two weeks prior to Period I doing.
10. Donating greater than 150 mL of blood within two months prior to Period I dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study.
11. Consumption of caffeine, xanthine-containing products (i.e. coffee, tea, caffeine-containing sodas, colas and chocolate, etc.) and/or alcohol, smoke or use tobacco products within 48 hours prior to days on which dosing is scheduled and during the periods when blood samples are being collected.
12. Any other medical reason as determined by the clinical investigator.
13. Subject is pregnant or breastfeeding.
14. Women of childbearing potential disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs): | 24 hours
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Pharmacokinetic profile of maximum concentration of HUYPS-1 (Cmax) | 24 hours
  Concentrations of HUYPS-1 and it metabolites in plasma and urine will be measured by a specific and sensitive LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  Cmax
Pharmacokinetic profile of time of occurrence for maximum (peak) HUYPS-1 concentration (Tmax) | 24 hours
  Concentrations of HUYPS-1 and it metabolites in plasma and urine will be measured by a specific and sensitive LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  Tmax
Pharmacokinetic profile of area under curve (AUC0-t) for HUYPS-1 | 24 hours
  Concentrations of HUYPS-1 and it metabolites in plasma and urine will be measured by a specific and sensitive LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  AUC0-t
Pharmacokinetic profile of area under curve infinity (AUCINF) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  AUCINF
Pharmacokinetic profile of overall HUYPS-1 elimination rate constant (k) | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  k
Pharmacokinetic profile of elimination half-life (T1/2) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  T1/2
Pharmacokinetic profile of mean residence time (MRT) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  MRT
Pharmacokinetic profile of clearance (CL/F) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  CL/F
Pharmacokinetic profile of apparent volume (Vd/F) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  Vd/F
Pharmacokinetic profile of area under moment curve (AUMC(0-t)) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  AUMC(0-t)
Pharmacokinetic profile of area under moment curve infinity (AUMCINF) for HUYPS-1 | 24 hours
  LC/MS/MS method developed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. According to the pharmacokinetic parameters of HUYPS-1 and its metabolites in health subjects oral HUYPS-1 to assess the safety information.The study will be conducted to validate the precision, accuracy (including with-run and between-run variation), linearity, specificity, reproducibility, limit of quantitation based on recovery studies. Assays will be performed in the laboratory of Clinical Pharmacokinetic Laboratory of Tri-Service General Hospital. Spiked samples of known concentrations will be analyzed together for quality control of the assay method.
  The following parameters of HUYPS-1 will be determined using WINNONLINTM:
  AUMCINF

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No